CLINICAL TRIAL: NCT02340780
Title: A Phase II Study of Buparlisib in Patients With Relapsed and Refractory Chronic Lymphocytic Leukemia
Brief Title: Buparlisib in Patients With Relapsed and Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I216
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2020-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buparlisib (Experimental): 100mg daily orally every 28 days
  Interventions: Drug: Buparlisib

INTERVENTIONS:
Drug: Buparlisib

SUMMARY:
The purpose of this study is to find out what effects a new drug, buparlisib, has on chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Buparlisib has been shown to shrink tumours in animals. It has been studied in some people and seems promising but it is not clear if it can offer better results than standard treatment.

The standard or usual treatment for this disease is chemotherapy, targeted therapy or radiation, either alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* Previously documented CLL that is recurrent or relapsed after previous therapy and that requires treatment
* Age ≥ 18 years
* ECOG Performance Status score of 0, 1 or 2
* Patients must have a life expectancy of at least 12 weeks. Those who have previously completed curative treatment of a malignancy other than CLL will be eligible
* Patients must have at least ONE of: Lymphocyte count ≥ 10 x 10^9/L OR at least one pathologically enlarged lymph node (≥ 2 x 2 cm) by CT scan
* Previous therapy: Patients must have received at least 1 prior systemic treatment regimen (single agent or combination therapy). There is no upper limit on number of prior regimens. Patients who have received prior autologous or allogeneic stem cell transplantation are eligible.
* Patients must have recovered (to ≤ grade 2) from all reversible toxicity related to prior systemic therapy, and have adequate washout from prior chemotherapy and investigational agents defined as the longest of:

  * two weeks
  * standard cycle length of prior regimen (e.g. 28 days for FCR)
  * 5 half-lives for investigational drugs

Not permitted:

• prior treatment with buparlisib (BKM120)

* Patients may have had radiation, provided a minimum of 21 days has elapsed prior to enrollment. Patients must have recovered from any acute toxic effects from radiation prior to registration
* Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed if surgery was major
* Absolute neutrophil counts (ANC): ≥ 1.0 x 10^9/L
* Platelets ≥ 50/min x 10^9/L and more than 5 days since last transfusion
* Creatinine clearance* ≥ 50 mL/min
* Bilirubin** ≤ 1.5 x upper normal limit (UNL)
* Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 1.5 x UNL or ≤ 3 x UNL if hepatic involvement with CLL
* Potassium and calcium Within normal limits for laboratory (supplementation permitted)
* Glucose (fasting) < 7.8 mmol/L (AND HbA1c ≤ 8% if diabetic)

  * Creatinine clearance as calculated by Cockcroft-Gault formula or by 24 hour urine measurement: Females: GFR = 1.04 x (140-age) x weight in kg serum creatinine in μmol/L Males: GFR = 1.23 x (140-age) x weight in kg serum creatinine in μmol/L

  ** Direct if patient known to have Gilbert's syndrome
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient registration

Exclusion Criteria:

* Progression to high grade lymphoma (Richter's transformation) or myelodysplasia
* Patients with known hypersensitivity to the study drug or its excipients
* The following are exclusions for enrolment on the study:

  * Pregnant or lactating women. (N.B. All women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration).
  * Men and women of childbearing potential who do not agree to use adequate contraception: prior to study entry; while taking buparlisib and after completion of study therapy for 12 weeks in men and 4 weeks in women.
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including, but not limited to:

  1. active uncontrolled or serious infection (viral, bacterial or fungal);
  2. pulmonary disease requiring oxygen;
  3. known HIV infection or other immune deficiency disorders (except for CLL);
  4. uncontrolled auto-immune hemolytic anemia (AIHA) or auto-immune thrombocytopenia (ITP)
  5. acute or chronic pancreatitis
* Uncontrolled or significant cardiovascular disease including:

  * Myocardial infarction within 12 months
  * Uncontrolled angina within 6 months
  * Clinically significant congestive heart failure (eligible if controlled and LVEF ≥ 50%)
  * Stroke, TIA or other ischemic event within 12 months
  * Severe cardiac valve dysfunction
  * Left ventricular ejection fraction < 50% (only required if symptoms suggestive or history of cardiovascular disease)
  * Uncontrolled hypertension
* Patient has any of the following mood disorders:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others)
  * Score of ≥ 12 on the PHQ-9 questionnaire
  * Score of ≥ 15 on the GAD-7 mood scale
  * ≥ CTCAE grade 3 anxiety
  * Patient selects a positive response of '1,2,3' to question 9 (suicidal ideation) in the PHQ-9 questionnaire
* Patients who have received prior buparlisib (BKM120).
* Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of buparlisib (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients who are unable to swallow capsules
* Patients on strong CYP3A inhibitors/inducers or therapeutic doses of warfarin-like anticoagulants (must have discontinued > 7 days prior to day 1). Patients may receive low molecular weight heparin if indicated. See Appendix VII for a list of prohibited medications.
* Patients on drugs with a known risk to induce Torsades de Pointes
* Patients receiving high dose steroid therapy or another immunosuppressive agent. Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients who are on stable moderate dose corticosteroid treatment for treatment of conditions other than CLL (< dexamethasone 4 mg/day, prednisone 25 mg/day) for at least 14 days before start of study treatment are eligible.
* Patients with known HIV positivity.
* Patients with known CLL involvement of the central nervous system.
* Patients with a history of other malignancies, except those which have been curatively treated and require no ongoing therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Assouline, Study Chair — McGill University - Dept. Oncology, Jewish General Hospital Site, Montreal QC Canada
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Assouline S, Amrein L, Aloyz R, Banerji V, Caplan S, Owen C, Hasegawa W, Robinson S, Shivakumar S, Prica A, Peters A, Hagerman L, Rodriguez L, Skamene T, Panasci L, Chen BE, Hay AE. IND.216: a phase II study of buparlisib and associated biomarkers, raptor and p70S6K, in patients with relapsed and refractory chronic lymphocytic leukemia. Leuk Lymphoma. 2020 Jul;61(7):1653-1659. doi: 10.1080/10428194.2020.1734594. Epub 2020 Mar 10. PMID 32154751

RESULTS

PARTICIPANT FLOW:
Groups:
- Buparlisib: 100mg daily orally every 28 days
  Buparlisib
Period: Overall Study
Arm/Group | Buparlisib
Started | 14 (A total of 14 patients enrolled, one patient was found ineligible after the enrollment.)
Completed | 13
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients will be included in the analysis.
Arm/Group | Buparlisib
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 74 [61 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Performance status [Count of Participants; unit: Participants] — The scale was developed by the Eastern Cooperative Oncology Group (ECOG)
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    Grade 0 | 5
    Grade 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate (complete + partial response, as defined in the protocol) to oral buparlisib in patients with relapsed and refractory chronic lymphocytic leukemia.
  Complete Response (CR): CR requires all of the criteria listed on page 31 of the protocol, maintained for a period of at least 8 weeks.
  Partial Response (PR): To define a PR, at least 1 of the criteria of Group A plus 1 of the criteria of Group B listed on page 32 of the protocol must be met and persist for ≥ 8 weeks, in the absence of any criteria definitive of progressive disease.
Time Frame: 30 months
Population: All eligible patients who received the protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Buparlisib
Number analyzed (Participants) | 13
Participants
  Response | 6
  Non-response | 7

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time in months from study entry until disease progression or death.
Time Frame: 30 months
Population: All eligible patients who received protocol treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Buparlisib
Number analyzed (Participants) | 13
months | 21.65 [5.36 to NA] — Due to small sample size and small number of events, the upper limit of the 95% confidence interval is not available.

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Buparlisib
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (N=13)
Nausea (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Other surgical and medical procedures (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (N=13)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Other ear and labyrinth disorders (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Other endocrine disorders (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 2
Cataract (Eye disorders) | 1
Other eye disorders (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Other gastrointestinal disorders (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 8
Fever (General disorders) | 1
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Other general disorders, administration site conditions (General disorders) | 2
Pain (General disorders) | 2
Lung infection (Infections and infestations) | 1
Other infections and infestations (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Other injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Other nervous system disorders (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Other psychiatric disorders (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Other surgical and medical procedures (Surgical and medical procedures) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Other vascular disorders (Vascular disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02340780/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02340780/SAP_000.pdf